## Exploring the role of tryptophan metabolites in pediatric migraine

## **Informed Consent Form**

Dear study participant, Hello, we hereby invite you to participate in a medical research project in which 200 participants are expected. This informed consent formprovides you with some information to help you decide whether to participate in this study. Please read the following carefully and discuss any questions or terms that areunclear with your study physician.

Background and purpose of the study: The overall prevalence of migraine in thepediatric population is approximately 7.7%, increasing from approximately 5% inchildhood to 15% in adolescence. Migraine is often associated with cerebrovasculardisease, epilepsy, and depression, and the effectiveness of medication for migraine isunclear, with a high recurrence rate, which seriously affects children's school life andphysical and mental health. This study will investigate the relationship between poorlifestyle and migraine attacks, compare the levels of serum markers of tryptophanmetabolites in children with migraine with those in healthy children, assess the impactof different prognostic factors on the prognosis of migraine in children, and urgeparents and children to change their lifestyle, reduce migraine drug dependence.improve migraine treatment and improve the prognosis.

**Methods:** Parents and children will fill out the questionnaire together and 5 ml ofelbow vein blood will be collected from the child. There may be risks of pain, bloodsickness, and dislodgement of the blood collection needle during the blood collectionprocess, but it generally does not cause significant prolonged discomfort to the child. No additional blood is collected for the study, and the samples collected are leftoverblood samples from normal visits and do not incur additional costs.

**Possible benefits:** The poor lifestyle of children with migraine can be investigated and parents and children can be urged to make lifestyle changes to improve theirhealth. Differences in serum markers between children with migraine and healthychildren can be detected to improve the diagnosis of migraine, predict the risk of migraine, improve the prognosis of children with migraine, and provide early relief of pain and improve quality of life.

Your Rights and Responsibilities: The executive arm of this clinical researchprogram will uphold your rights and interests during the course of the study. Yourmedical records (e.g., test results, physician's diagnosis) will be kept confidential bythe investigators and coding will be used in place of your name. Data from the studymay be published for academic purposes, but your privacy (e.g, name, cell phonenumber, etc.) will not be disclosed, You can stay informed about the information andresearch progress related to this study, and if you have any questions during the study.please contact Junhui Liu, whose contact number is 15064039296.

I have read the above information, I have had the opportunity to ask relevant

questions and my questions have been answered to my satisfaction. I voluntarily agreeto participate in this study as a subject and understand that I have the right towithdraw from this study at any time without in any way affecting my future medicatreatment.

**Signature of subject:** Signature of guardian:Date:I have fully explained to the subject (name). The subject of the investigation hassufficient knowledge of this study.

| Signature of subject: |
|------------------------|
| Signature of guardian: |
| Date: |